CLINICAL TRIAL: NCT04532086
Title: Relationship Between Uterocervical Angle and Prediction of Spontaneous Preterm Birth
Brief Title: Uterocervical Angle and Preterm Labour
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohammed Shaaban Abd Al Razik Ibrahim, Principal investigator, Ain Shams Maternity Hospital
Other Study IDs: UCA in preterm birth
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Preterm Labor
Keywords: uterocervical angle; Preterm birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Uterocervical angle — Transvaginal ultrasound examination will be performed at 18-28 weeks gestation in (197) pregnant women with live singleton fetuses, attending routine prenatal care services. Measuring length of uterine cervix at (18-28) weeks & evaluation of dilatation of internal os & measurement of uterocervical angle between(18-28)weeks gestational age.

SUMMARY:
To determine whether a novel ultrasonographic marker, uterocervical angle, correlates with risk of spontaneous preterm birth

DETAILED DESCRIPTION:
The uterocervical angle is the triangular segment measured between the lower uterine segment and the cervical canal, yielding a measurable angle. The first ray was placed from the internal os to the external os. The calipers were placed where the anterior and posterior walls of the cervix touch the internal and external os along the endocervical canal. If the cervix was curved, the first ray was also drawn from the internal os to the external os as a straight line. A second ray was then drawn to delineate the lower uterine segment. This ray was traced up the anterior uterine segment to a distance allowed by the preloaded image. Ideally, the second ray would reach 3cm up the lower uterine segment in order to establish an adequate measurement. The anterior angle in between the two rays was measured with a protractor. In the presence of funneling, the first ray was placed to measure the length of remaining cervix. The second caliper was placed from the innermost portion of measurable cervix and extended to the lower uterine segment. In the event that the lower uterine segment was found to be irregular, the second caliper was placed centrally along the segment. In the event of a retroverted uterus, the angle should be measured in a similar fashion with the first ray along the measurable cervix and the second ray traced along the lower uterine segment. Unlike in an anteverted or axial positioned uterus, however, the posterior side of the angle closer to the intrauterine contents should then be measured.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age (18_40).
* BMI (20_34).
* singleton gestations between (18 - 28) weeks.
* Multiparity.
* History of previous preterm deliveries or mid-trimesteric abortions.

Exclusion Criteria:

* Loss of follow up.
* Preterm premature rupture of membranes(PPROM).
* Placental abnormalities.
* Past history of cervical operations.
* Multifetal pregnancy.
* Polyhydramnios.
* Steroids intake .
* Medically or obstetric indicated pregnancy termination.
* Serious maternal or fetal problems.
* Cerclage during current pregnancy before the screening.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 197 pregnant women with singleton gestations between (18 - 28) weeks with history of previous preterm deliveries or mid-trimesteric abortions.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Gestational age at birth | 6 months
  Preterm labour is defined as regular contractions of the uterus resulting in changes in the cervix that start before 37 weeks of pregnancy. Changes in the cervix include effacement (the cervix thins out) and dilation (the cervix opens so that the fetus can enter the birth canal).

SECONDARY OUTCOMES:
Apgar score at 1 and 5 minutes | 6 months
  Appearance (skin color) Pulse (heart rate) Grimace response (reflexes) Activity (muscle tone) Respiration (breathing rate and effort)

CONTACTS AND LOCATIONS:
Overall Officials: Osama Is Kamel, lecturer, Study Director — Lecturer; Wessam Mg Abuelghar, Professor, Study Director — Professor; Ahmed Kh Makled, Professor, Study Director — Professor

REFERENCES:
- [Background] Daskalakis G, Theodora M, Antsaklis P, Sindos M, Grigoriadis T, Antsaklis A, Papantoniou N, Loutradis D, Pergialiotis V. Assessment of Uterocervical Angle Width as a Predictive Factor of Preterm Birth: A Systematic Review of the Literature. Biomed Res Int. 2018 Dec 26;2018:1837478. doi: 10.1155/2018/1837478. eCollection 2018. PMID 30687736
- [Background] Swanson K, Grobman WA, Miller ES. Is Uterocervical Angle Associated with Gestational Latency after Physical Exam Indicated Cerclage? Am J Perinatol. 2018 Jul;35(9):840-843. doi: 10.1055/s-0037-1621734. Epub 2018 Jan 24. PMID 29365330
- [Background] van der Merwe J, Couck I, Russo F, Burgos-Artizzu XP, Deprest J, Palacio M, Lewi L. The Predictive Value of the Cervical Consistency Index to Predict Spontaneous Preterm Birth in Asymptomatic Twin Pregnancies at the Second-Trimester Ultrasound Scan: A Prospective Cohort Study. J Clin Med. 2020 Jun 8;9(6):1784. doi: 10.3390/jcm9061784. PMID 32521741
- [Background] Oskovi Kaplan ZA, Ozgu-Erdinc AS. Prediction of Preterm Birth: Maternal Characteristics, Ultrasound Markers, and Biomarkers: An Updated Overview. J Pregnancy. 2018 Oct 10;2018:8367571. doi: 10.1155/2018/8367571. eCollection 2018. PMID 30405914